CLINICAL TRIAL: NCT07371650
Title: A Multicenter, Open-Label, Randomized Phase 2a Study to Evaluate the Safety and Efficacy of Different Oral Doses of TRX-100 and Standard of Care in Participants With Influenza
Brief Title: This is an Early-stage Clinical Trial to Determine a Safe and Effective Dose for Tivoxavir Marboxil in Patients With Mild to Moderate Influenza
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRX-100-0002
Record Dates: First submitted 2025-08-04; First posted 2026-01-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 3 study arms (30 participant per arm) to receive study drug and standard of care therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRX-100 Dose Level 1 (Experimental): Participants in this arm will receive a lower single oral dose of the investigational drug, TRX-100.
  Interventions: Drug: TRX-100
- TRX-100 Dose Level 2 (Experimental): Participants in this arm will receive a higher single oral dose of the investigational drug, TRX-100.
  Interventions: Drug: TRX-100
- Standard of Care (SOC) (Active Comparator): Participants in this arm will not receive the investigational drug. Instead, they will receive the current standard of care treatment. This arm serves as a comparator to evaluate the effects of the investigational drug.
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: TRX-100 — CEN inhibitor, dosage form - capsules, dosing regimen - QD
  Arms: TRX-100 Dose Level 1; TRX-100 Dose Level 2
Drug: Standard of Care (SOC) — Standard of Care Influenza Antiviral therapy
  Arms: Standard of Care (SOC)

SUMMARY:
This is an early-stage clinical trial to determine a safe and effective dose for Tivoxavir Marboxil (TRX-100) in patients with mild to moderate Influenza. Participants will take a study drug as well as a standard therapy. A descriptive statistics will be used to present the study results.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, Phase 2a study to evaluate the safety, tolerability, and pilot efficacy of different oral doses of TRX-100 in otherwise healthy participants with mild to moderate influenza. The study will also evaluate PK of TRX-100 and its major active metabolite, TRX-101, following single oral doses of TRX-100.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of influenza A or B virus infection
* The time interval between the onset of symptoms and enrollment is 48 hours or less
* Satisfactory baseline medical assessment by history and physical examination

Exclusion Criteria:

* Positive test results for SARS-CoV-2 infection and/or respiratory syncytial virus infection
* Participants with concurrent infections requiring systemic antimicrobial therapy
* Participants with any serious or chronic underlying disease likely to affect study outcomes at the Investigator's discretion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE | up to Day 28
  Number of participants with Adverse Events (AEs), serious Adverse Events (SAEs) (including withdrawals due to AEs)
Incidence of abnormal laboratory tests results | Up to Day 28
  Number of participants with abnormal laboratory tests results
Incidence of abnormal clinically significant ECG results | Up to 28 days
Number of participants with abnormal physical examinations findings | Up to 28 days

SECONDARY OUTCOMES:
Change from baseline in the total score of 7 influenza symptoms | up to Day 15
  Seven symptoms (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, and fatigue) will be assessed by the participant and recorded on a 4-point severity scale
Plasma Tmax | PK samples will be collected from Day 1 through Day 22.
  Time to reach the maximum plasma concentration of TRX-100.
Incidence of influenza-related complications | Up to 28 days
Time to alleviation of influenza clinical symptoms (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, and fatigue) | Up to 28 days
Time to resolution of fever to <37 C (axillary temperature) | Up to 28 days
Percentage of participants with resolution of fever | Up to 28 days
Time needed to return to pre-influenza health status based on assessment of activities score | Up to 28 Days
Plasma Cmax | PK samples will be collected from Day 1 through Day 22.
  TRX-100 peak plasma concentration
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of TRX-100 | PK samples will be collected from Day 1 through Day 22.
Plasma Cmax | PK samples will be collected from Day 1 through Day 22.
  TRX-101 peak plasma concentration
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of TRX-101 | PK samples will be collected from Day 1 through Day 22.
Area under the plasma concentration-time curve from time zero to 24 hours post-dose (AUC0-24) | PK samples will be collected from Day 1 through Day 22.
  Area under the plasma concentration-time curve from time zero to 24 hours post-dose for TRX-100.
Area under the plasma concentration-time curve from time zero to 24 hours post-dose (AUC0-24) | PK samples will be collected from Day through Day 22
  Area under the plasma concentration-time curve from time zero to 24 hours post-dose for TRX-101.
Area under the plasma concentration-time curve from time zero extrapolated to infinity | PK samples will be collected from Day 1 through Day 22.
  A measure of total drug exposure from administration extrapolated to infinite time, estimated for TRX-100.
Area under the concentration-time curve extrapolated to infinity | PK samples will be collected from Day 1 through Day 22.
  A measure of total drug exposure from administration extrapolated to infinite time, estimated for TRX-101.
Terminal elimination half-life | PK samples will be collected from Day 1 through Day 22.
  The time required for the plasma concentration of TRX-100 to decrease by 50% in the terminal elimination phase.
Terminal elimination half-life | PK samples will be collected from Day 1 through Day 22
  The time required for the plasma concentration of TRX-101 to decrease by 50% in the terminal elimination phase.
Terminal elimination rate constant | PK samples will be collected from Day 1 through Day 22
  The first-order rate constant associated with the terminal elimination phase of the plasma concentration-time curve for TRX-100.
Terminal elimination rate constant. | PK samples will be collected from Day 1 through Day 22
  The first-order rate constant associated with the terminal elimination phase of the plasma concentration-time curve for TRX-101.
Apparent oral clearance (CL/F) | PK samples will be collected from Day 1 through Day 22
  Apparent total clearance of TRX-100 from plasma following oral administration
Apparent oral clearance (CL/F) | PK samples will be collected from Day 1 through Day 22
  Apparent total clearance of TRX-101 from plasma following oral administration
Apparent volume of distribution during the terminal phase | PK samples will be collected from Day 1 through Day 22.
  Apparent volume of distribution of TRX-100 during the terminal elimination phase following oral administration, calculated as Clearance (CL/F) divided by the elimination rate constant.
Apparent volume of distribution during the terminal phase | PK samples will be collected from Day 1 through Day 22.
  Apparent volume of distribution of TRX-101 during the terminal elimination phase following oral administration, calculated as Clearance (CL/F) divided by the elimination rate constant.
Plasma Tmax | Time Frame: PK samples will be collected from Day 1 through Day 22.
  Time to reach the maximum plasma concentration of TRX-101.
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of TRX-101. | PK samples will be collected from Day 1 through Day 22.

OTHER OUTCOMES:
Change from Baseline in Viral Titer | up to Day 6
  Change of virus titer compared to pretreatment baseline sample
Change from Baseline in Viral Load | up to Day 6
  Change in virus load compared to pretreatment baseline sample

CONTACTS AND LOCATIONS:
Locations (1):
- Novatrials, Charlestown, New South Wales, Australia